CLINICAL TRIAL: NCT01768429
Title: The Effect of n-3 Fatty Acids and Fish on Glucose and Lipid Metabolism in Subjects With Impaired Glucose Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other); VTT Technical Research Centre, Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: ALFAKALA
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Hyperglycemia
MeSH Terms: conditions — Hyperglycemia | interventions — bearberry, bladderwrack, borage oil, centella, fatty acid, fish oil, ginkgo biloba, melilotus, soya lecithin drug combination; alpha-Linolenic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fatty fish (Experimental): Four fatty fish meals per week
  Interventions: Behavioral: Fatty fish
- Lean Fish (Experimental): Four lean fish meals per week
  Interventions: Behavioral: Lean Fish
- Alpha-linolenic acid (Experimental): 10 g of alpha-linolenic acid daily from camelina sativa oil
  Interventions: Behavioral: Alpha-linolenic acid
- Control diet (Experimental): Limited fish and alpha-linolenic acid intake
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Fatty fish
  Arms: Fatty fish
Behavioral: Lean Fish
  Arms: Lean Fish
Behavioral: Alpha-linolenic acid
  Arms: Alpha-linolenic acid
Behavioral: Control
  Arms: Control diet

SUMMARY:
The aim of the project is to examine whether the sources of n-3 fatty acids and fish itself differ in their effects on glucose metabolism, lipid metabolism, blood pressure, and serum inflammatory markers. Lipidomic profiles and gene expression will be used for thorough assessment of the possible clinical changes. The study will compare the effects of alpha-linolenic acid containing vegetable oil, fatty fish, lean fish and control diet. The results of this project will help to identify the optimal source of n-3 fatty acids, and reveal the significance of the components of fish other than fatty acids. These data will be useful both nationally and internationally, since highly controlled dietary interventions utilizing new methodology are scarce.

ELIGIBILITY:
Inclusion Criteria:

* age 40-70 years
* BMI 25-32 kg/m2
* fasting plasma glucose 5.6-7.0 mmol/l
* 2 h plasma glucose in oral glucose tolerance test <=11 mmol/l
* fasting serum total cholesterol <=7 mmol/l
* fasting serum LDL cholesterol <=5 mmol/l
* fasting serum triglycerides <=4 mmol/l

Exclusion Criteria:

* any chronic disease or condition that hamper the ability to follow dietary intervention
* chronic liver, thyroid or kidney disease
* alcohol abuse
* diabetes
* recent weight loss
* recent myocardial infarction
* corticosteroid therapy
* psychiatric disorders which need drug treatment
* cancer under treatment
* fish allergy or other extensive food allergies
* exceptional diets (like Atkin's or vegan diet)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism assessed by oral glucose tolerance test and frequently sampled intravenous glucose tolerance test | Baseline and 12 weeks
  change in glucose metabolism
Serum lipid profile | Baseline and at 12 weeks
  Change in serum lipid profile
Blood pressure | Baseline and 12 weeks
  Change in blood pressure
Serum inflammatory markers | baseline and 12 weeks
  Change in serum inflammatory markers
Plasma and adipose tissue lipidomic profile | Baseline and 12 weeks
  Change in plasma and adipose tissue lipidomic profile
Plasma and urine metabonomics | Baseline and 12 weeks
  Change in plasma and urine metabonomics
Gene expression in adipose tissue and peripheral blood mononuclear cells | Baseline and 12 weeks
  Change in gene expression in adipose tissue and peripheral blood mononuclear cells

SECONDARY OUTCOMES:
Reverse cholesterol transport | Baseline and 12 weeks
  Change in reverse cholesterol transport

CONTACTS AND LOCATIONS:
Overall Officials: Arja Erkkilä, Adjunct Prof, Principal Investigator — University of Eastern Finland; Ursula Schwab, Adjunct Prof, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio, Finland

REFERENCES:
- [Derived] Meuronen T, Lankinen MA, Fauland A, Shimizu BI, de Mello VD, Laaksonen DE, Wheelock CE, Erkkila AT, Schwab US. Intake of Camelina Sativa Oil and Fatty Fish Alter the Plasma Lipid Mediator Profile in Subjects with Impaired Glucose Metabolism - A Randomized Controlled Trial. Prostaglandins Leukot Essent Fatty Acids. 2020 Aug;159:102143. doi: 10.1016/j.plefa.2020.102143. Epub 2020 May 30. PMID 32512364
- [Derived] Manninen S, Lankinen M, Erkkila A, Nguyen SD, Ruuth M, de Mello V, Oorni K, Schwab U. The effect of intakes of fish and Camelina sativa oil on atherogenic and anti-atherogenic functions of LDL and HDL particles: A randomized controlled trial. Atherosclerosis. 2019 Feb;281:56-61. doi: 10.1016/j.atherosclerosis.2018.12.017. Epub 2018 Dec 23. PMID 30658192
- [Derived] Manninen S, Lankinen M, de Mello V, Agren J, Laaksonen D, Schwab U, Erkkila A. The effect of camelina sativa oil and fish intakes on fatty acid compositions of blood lipid fractions. Nutr Metab Cardiovasc Dis. 2019 Jan;29(1):51-61. doi: 10.1016/j.numecd.2018.10.002. Epub 2018 Oct 11. PMID 30454883
- [Derived] Manninen SM, Lankinen MA, de Mello VD, Laaksonen DE, Schwab US, Erkkila AT. Intake of Fatty Fish Alters the Size and the Concentration of Lipid Components of HDL Particles and Camelina Sativa Oil Decreases IDL Particle Concentration in Subjects with Impaired Glucose Metabolism. Mol Nutr Food Res. 2018 May;62(10):e1701042. doi: 10.1002/mnfr.201701042. PMID 29645359